CLINICAL TRIAL: NCT01298557
Title: Magnetoencephalography and High-Field Diffusion Tensor Magnetic Resonance Imaging of Neural Function and Connectivity in Traumatic Brain Injury
Brief Title: MEG and DTI of Neural Function and Connectivity in Traumatic Brain Injury
Acronym: Dana-REAC
Status: Completed | Type: Observational
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Other Study IDs: Dana-REAC
Record Dates: First submitted 2011-02-09; First posted 2011-02-17 (Estimated); Last update posted 2018-12-04 (Actual); Status verified 2018-11

CONDITIONS: Traumatic Brain Injury; Post-concussive Symptoms
Keywords: Traumatic brain injury; Post-concussive symptoms; Brain imaging; Neurocognitive testing
MeSH Terms: conditions — Brain Injuries, Traumatic; Post-Concussion Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Traumatic brain injured patients: This group consists of participants who suffered a traumatic brain injury an average of 4 months to 4 years prior to testing. Patients must not have history of prior head injury, substance abuse, psychiatric illness, or contraindications to MRI.
- Controls (no traumatic brain injury): This group consists of participants who do not have a history of brain trauma. Furthermore, controls must not suffer from substance abuse, psychiatric illness, or have contraindications to the MRI.

SUMMARY:
The overall hypothesis is that the long-term cognitive and behavioral sequelae of traumatic brain injury (TBI) are due to selective disruption of the long association white matter tracts of the cerebral hemispheres, with resulting functional impairment of the network of cortical regions that are interconnected by these long-range association pathways. We propose that traumatic white matter injury can be measured with diffusion tensor imaging (DTI) and that the impaired cortical activation can be detected with magnetoencephalography (MEG), and that the results of these imaging examinations will correlate with neurocognitive status and functional recovery after TBI.

ELIGIBILITY:
Inclusion Criteria:

* 18-50 years of age
* single episode of blunt traumatic brain injury
* symptoms of persistent post-concussive syndrome present an average of 4 months to 4 years since date of injury
* fluency in English (cognitive battery not available in other languages)
* capable of self-consent

Exclusion Criteria:

* < 18 years or > 50 years of age
* pregnancy
* history of previous TBI with loss of consciousness
* alcoholism as evidenced by Audit questionnaire
* regular use of illicit drugs
* non-English fluency
* significant psychiatric history excluding mild depression or anxiety disorder any contraindication to MRI, including claustrophobia, pregnancy, any trauma or surgery which may have left ferromagnetic material in the body, ferromagnetic implants or pacemakers; and inability to lie still for 1 hour or more

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Participants will be recruited through the neurosurgery clinic at San Francisco General Hospital or referred to us by colleagues.
Sampling Method: Non-Probability Sample
Enrollment: 69 (Actual)
Dates: Start 2007-02; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Changes in white matter tract structure | up to 4 years following date of injury
  We believe that brain injury results in selective disruption of the associative white matter tracts of the cerebral hemispheres, with resulting functional impairment of the network of cortical regions that are interconnected by these long-range association pathways. We propose that traumatic white matter injury can be measured with diffusion tensor imaging (DTI). We evaluate DTI using 3T and 7T MRI. Participants receive scans at only one time-point.

SECONDARY OUTCOMES:
Neurocognitive function | up to 4 years following date of injury
  We hope to better understand the long-term cognitive and behavioral sequelae of traumatic brain injury (TBI) by correlating neurocognitive testing data with imaging data. We will also compare neurocognitive testing data between patients and controls to help illustrate the impact of brain trauma on these neurocognitive symptoms. Our participants receive testing at only one time-point.
Cortical activation | up to 4 years following date of injury
  We believe that brain injury results in selective disruption of the associative white matter tracts of the cerebral hemispheres, with resulting functional impairment of the network of cortical regions that are interconnected by these long-range association pathways. We propose that impaired cortical activation can be detected with magnetoencephalography (MEG). We will compare patients' data with data of controls. Our participants are scanned at only one time-point.

CONTACTS AND LOCATIONS:
Overall Officials: Pratik Mukherjee, MD, PhD, Principal Investigator — UCSF Department of Radiology and Bioengineering
Locations (1):
- San Francisco General Hospital, San Francisco, California, United States

REFERENCES:
- [Background] Arfanakis K, Haughton VM, Carew JD, Rogers BP, Dempsey RJ, Meyerand ME. Diffusion tensor MR imaging in diffuse axonal injury. AJNR Am J Neuroradiol. 2002 May;23(5):794-802. PMID 12006280
- [Background] Deipolyi AR, Mukherjee P, Gill K, Henry RG, Partridge SC, Veeraraghavan S, Jin H, Lu Y, Miller SP, Ferriero DM, Vigneron DB, Barkovich AJ. Comparing microstructural and macrostructural development of the cerebral cortex in premature newborns: diffusion tensor imaging versus cortical gyration. Neuroimage. 2005 Sep;27(3):579-86. doi: 10.1016/j.neuroimage.2005.04.027. PMID 15921934
- [Background] Hillebrand A, Singh KD, Holliday IE, Furlong PL, Barnes GR. A new approach to neuroimaging with magnetoencephalography. Hum Brain Mapp. 2005 Jun;25(2):199-211. doi: 10.1002/hbm.20102. PMID 15846771
- [Background] Hughes DG, Jackson A, Mason DL, Berry E, Hollis S, Yates DW. Abnormalities on magnetic resonance imaging seen acutely following mild traumatic brain injury: correlation with neuropsychological tests and delayed recovery. Neuroradiology. 2004 Jul;46(7):550-8. doi: 10.1007/s00234-004-1227-x. Epub 2004 Jun 8. PMID 15185054
- [Background] Huisman TA, Sorensen AG, Hergan K, Gonzalez RG, Schaefer PW. Diffusion-weighted imaging for the evaluation of diffuse axonal injury in closed head injury. J Comput Assist Tomogr. 2003 Jan-Feb;27(1):5-11. doi: 10.1097/00004728-200301000-00002. PMID 12544235